CLINICAL TRIAL: NCT00170144
Title: Branched Chain Amino Acids as Stimulant of Muscle Mitochondrial Function in Elderly People
Brief Title: Effect of Branched Chain Amino Acids on Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 05-004000
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
MeSH Terms: interventions — Amino Acids

INTERVENTIONS:
Drug: Branchamin 4%

SUMMARY:
With aging, there is a decrease in muscle mass and function especially in the energy storehouses of cells called mitochondria. Amino acids, the building blocks of protein, and insulin have been shown to increase muscle mitochondrial protein synthesis and thereby function. Branched chain amino acids which can only be provided in the diet seem to be key in this process. Therefore in our study, our aim is to study the effect of branched chain amino acids on muscle mitochondrial protein synthesis in both the young and elderly. By doing so, we can then elucidate if branched chain amino acid supplementation has future potential in improving quality of life and performance in the elderly. The study will involve blood sampling and needle muscle biopsy.

DETAILED DESCRIPTION:
Skeletal muscle mito ATP production in young people are stimulated by insulin when infused with a mixture of amino acids while clamping blood glucose at the basal level. Our preliminary results indicate that this effect on mito ATP production is directly related to amino acid levels. Recent publications indicated that infusion of insulin with amino acids specifically stimulate muscle mitochondrial protein synthesis with no effect on synthesis or contractile proteins or sarcoplasmic proteins. The recent publications also indicated that intracellular amino acid anabolic sensors are stimulated by amino acids. It appears that BCAA, especially leucine has a specific effect in stimulating intracellular signaling or translation of mRNA to protein synthesis. It has been shown that amino acids, especially leucine, stimulate protein synthesis by activation of the mTOR pathway in mTOR phosphorylates p70S6 kinase which in turn phosphorylates the ribosomal S6 protein, resulting in increased activity of the protein synthesis complex. Activated mTOR also phosphorylates eIF4E-BP1 and activates the protein synthesis initiation complex. It is the abundance of specific mRNAase that determines synthesis of which specific proteins are promoted. Our preliminary data supports that amino acids selectively promotes muscle mitochondrial protein synthesis by enhancing the abundance of transcripts of genes that encode mitochondrial proteins. Administration of an amino acid mixture, specifically BCAA, is proposed as a stimulant of muscle mitochondrial ATP production. Secondary measurements will be performed to understand the underlying mechanism of enhanced muscle ATP production. These results are likely to contribute to our understanding of the basic mechanisms of the regulation of mitochondrial biogenesis in humans which will have potential future application.

This is a cross-sectional study between young and old. The study will use the new proteomic techniques established in our laboratory to profile and quantify mitochondrial protein synthesis in the participants. The combination of metabolic labeling with stable isotope and measuring synthesis rates of specific mito proteins by tandem mass spectrometry will determine whether actual stimulation by BCAA occurs differentially in young and elderly.

ELIGIBILITY:
Young (age 18-30) or old (age 65-80) Body mass index <30

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Does branched chain amino acids stimulate muscle mitochondrial ATP production in young and elderly?

SECONDARY OUTCOMES:
Does branched chain amino acids increase abundance of mRNA of genes encoding mitochondrial proteins and transcription factors equally in young and old?
Does branched chain amino acids increase levels of phosphorylated signaling proteins through the mTOR pathways equally in the young and old?
Does branched chain amino acids increase fractional synthesis rates of specific mitochondrial proteins, mitochondrial protein concentrations and mitochondrial enzyme activities equally in the young and old?

CONTACTS AND LOCATIONS:
Overall Officials: K. Sreekumaran Nair, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States